CLINICAL TRIAL: NCT06124690
Title: Persistent Atrial Fibrillation Without the Evidence of Low-voltage Areas: a Prospective Randomized Trial
Brief Title: Persistent Atrial Fibrillation Without the Evidence of Low-voltage Areas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Cathrin Theis, Principal Invetsigator, Head of Electrophysiology, Robert Bosch Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stuttgart, EP-004
Record Dates: First submitted 2023-09-26; First posted 2023-11-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Persistent Atrial Fibrillation; Catheter Ablation; Low Voltage Areas
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Patients with persistent atrial fibrillation are included in the study. They are randomized into three diffrenet treatment arms depending on the presence of left atrial fibrosis.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary vein isolation (no low voltage) (Active Comparator): Patients without the presence of low voltage areas receive pulmonary vein isolation only.
  Interventions: Device: Catheter ablation
- Pulmonary vein isolation only (evidence of low voltage areas) (Active Comparator): Patients with the evidence of low voltage areas are randomized to either pulmonary vein isolation only or PVI plus ablation of low voltage areas.
  Interventions: Device: Catheter ablation
- Pulmonary vein isolation plus ablation of low voltage areas (Active Comparator): Patients with the evidence of low voltage areas are randomized to either pulmonary vein isolation only or PVI plus ablation of low voltage areas.
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: Catheter ablation — Pulmonary vein isolation and ablation of low voltage areas.

SUMMARY:
An effective therapy of persistent atrial fibrillation beyond pulmonary vein isolation remains unsatisfactory. Targeting endocardial low-voltage areas represents an approach of substrate modification.

This prospective, randomized study investigated the efficacy of ablation of low-voltage areas versus PVI and additional linear ablations in patients with persistent atrial fibrillation in terms of single-procedure arrhythmia-free outcome and safety.

DETAILED DESCRIPTION:
Pulmonary vein isolation has become the cornerstone of the interventional treatment of paroxysmal atrial fibrillation. For the treatment of persistent atrial fibrillation the data remains unclear. All different approaches remain unsatisfactory for the treatment of persistent atrial fibrillation, including single pulmonary vein isolation, targeting endocardial areas of low-voltage, identifying areas with complex fractionated atrial electrograms (CFAE), ablating linear lines such as an anterior line, a roof-line or mitral isthmus line. Recurrence rates are still higher as compared to paroxysmal atrial fibrillation ablation. Several studies showed a good correlation between the volume of low-voltage areas (LVA) and the burden of atrial fibrillation. Earlier studies that investigated ablation therapy using a substrate-guided ablation as compared to circumferential pulmonary vein isolation (CPVI) alone, mostly showed no significant difference in recurrence rates between both approaches. In contrast, some other studies showed better outcomes when targeting low-voltage areas. However, there was significant heterogeneity in patient selection, mapping and ablation strategies and therefore, comparisons are hard to make.

The patients are randomized into three different treatment arms (Group 1: PVI alone if no low voltage areas are detected, Group 2: PVI alone if low voltage areas are detected, Group 3: PVI plus ablation of low voltage areas.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation according to the current guidelines
* Age > 18 years
* Patient information

Exclusion Criteria:

* Minors

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with atrial arrhythmia recurrence after 12 months follow-up | 12 months
  Number of participants with atrial arrhythmia recurrence after 12 months follow-up

SECONDARY OUTCOMES:
Number of procedural complications | 12 months
  Number of procedural complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Bosch Health Coampus, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No